CLINICAL TRIAL: NCT01252173
Title: MEASUREMENT OF ENDOTRACHEAL TUBE CUFF PRESSURE IN EMERGENCY DEPARTMENT PATIENTS
Status: Withdrawn | Type: Observational
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 120-05
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Intubation, Intratracheal
Keywords: endotracheal; intubation; tracheal; pressure; cufflator

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this research is to measure the endotracheal tube cuff pressure in patients who have been endotracheally intubated emergently in the emergency department or in the field by prehospital personnel. Overinflation of ETTc pressure is associated with injury, and we seek to determine if the phenomenon of excessively inflated ETTc can be detected in endotracheally intubated patients in the ED.

There is no experimental aspect to this study, it is only descriptive. Measurement of ETTc pressure is already performed by respiratory therapy/respiratory care. We simply seek to assess these measurements to determine if any patients in fact have high ETTc pressure. If it is found that patients do have ETTc with high pressures, this might allow emergency department staff or prehospital personnel such as paramedics or EMTs to use this information to seek methods by which endotracheal intubation can be improved and patients can be intubated without excessive ETTc pressure.

This is a pilot study. We have conducted several in vitro studies, which have all demonstrated that paramedics, EMTs, and emergency department physicians practice endotracheal intubation in a method that might result in excessively inflated ETTc.

ELIGIBILITY:
Inclusion Criteria:

* Patient emergently endotracheally intubated with a cuffed endotracheal tube.

Exclusion Criteria:

* Endotracheal intubation procedure performed in a setting other than the prehospital (field) or emergency department of participating institution. This specifically excludes endotracheally intubated patients transferred from another hospital, chronic care facility, or other location.
* Non-emergent or elective endotracheal intubation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All emergency department patients, and all patients admitted from the ED
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hoffman, MD, Principal Investigator — Beth Israel Medical Center